CLINICAL TRIAL: NCT05635071
Title: Prospective Clinical Study of Nintedanib to Inhibit Endometrial Fibrosis to Prevent Recurrence of Uterine Adhesions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022ZSLYEC-492
Record Dates: First submitted 2022-11-01; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Uterine Adhesions
Keywords: uterine adhesions; endometrail fibrisis
MeSH Terms: conditions — Gynatresia | interventions — nintedanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintedanib 100mg (Experimental): Traditional hormone replacement (HRT) cycle medication (Tegretol 2mg bid for 20 days, followed by Darvon 10mg bid for the last 10 days) + Nintedanib 100mg bid *15 days orally.
  Interventions: Drug: Nintedanib 100 MG [Ofev]
- Nintedanib 150mg (Experimental): Traditional hormone replacement (HRT) cycle medication (Tegretol 2mg bid for 20 days, followed by Darvon 10mg bid for the last 10 days) + Nintedanib 150mg bid *15 days orally.
  Interventions: Drug: Nintedanib 150 MG [Ofev]

INTERVENTIONS:
Drug: Nintedanib 100 MG [Ofev] — Nintedanib 100mg bid *15 days orally after hysteroscopic surgery
  Other Names: Nintedanib 100 MG Oral Capsule
  Arms: Nintedanib 100mg
Drug: Nintedanib 150 MG [Ofev] — Nintedanib 150mg bid *15 days orally after hysteroscopic surgery
  Other Names: Nintedanib 150 MG Oral Capsule
  Arms: Nintedanib 150mg

SUMMARY:
In moderate to severe cavity adhesions, the endometrial basal layer is more severely damaged and the regenerative capacity of the endometrium and glands is low. Even though hysteroscopic electrosurgery can roughly restore the cavity morphology, the postoperative recurrence rate is as high as 40%. Abnormal uterine cavity morphology and poor endometrial repair often lead to repeated cancellation of embryo transfer cycles in assisted reproduction treatment, and reduced clinical pregnancy rate, causing mental stress and financial burden to patients, which is one of the current problems in clinically assisted reproduction treatment. Nintedanib is a triple vascular kinase inhibitor that acts primarily on platelet-derived growth factor receptor (PDGFR) and fibroblast growth factor receptor (FGFR) and has been approved by the FDA for the clinical treatment of idiopathic pulmonary fibrosis and systemic sclerosis. The investigator's preliminary animal study found that endometrial fibrosis was significantly reduced in mice with gastric feeding of nintedanib in uterine adhesion molds. This study aimed to clarify further the role of nintedanib in inhibiting endometrial fibrosis and its clinical application value.

DETAILED DESCRIPTION:
The experiment will be divided into two groups based on the dose administered. After hysteroscopic surgery, one group will be given Nedanib 100mg bid orally for 15 days and the other group will be given Nedanib 150mg bid orally for 15 days. Hysteroscopic AFS scores and endometrial tissues before and after treatment will be collected for molecular biology experiments.

ELIGIBILITY:
Inclusion Criteria:

1)Clinical diagnosis of uterine adhesions; 2)Body mass index between 18-27 kg/m2; 3)Have a regular menstrual cycle of 27-35 days for at least six months; 4)Hysteroscopic diagnosis of moderate to severe uterine adhesions (AFS score >5), treated with electrodesiccation; 5)No contraindications to oral estrogen and progestin such as a history of thrombosis/breast tumor/history of abnormal liver function/migraine; 6)≥ 2 oocytes or blastocysts have been frozen.

Exclusion Criteria:

1)Patients with combined ovarian cysts ≥ 20 mm in diameter, submucosal uterine fibroids or intermuscular fibroids > 30 mm in diameter, pituitary tumors, and malignant tumors of various tissues and organs; 2)Patients with clinically significant abnormalities of the uterus (endometrial polyps, uterine malformations, endometriosis) and adnexa (hydrosalpinx); 3)Repeated implantation failures, such as three consecutive transfers with ≥6 failed high-quality embryos; 4)Known malformations of the reproductive organs that are unsuitable for pregnancy; 5)Abnormal cervical cytology (TCT) findings within 1 year before the screening; 6)Severe liver or kidney impairment, heart disease, or hypertension; 7)Known previous or current history of thrombophlebitis or thromboembolic disease; 8)Any known clinically significant systemic disease (e.g., diabetes mellitus, tuberculosis, etc; 9)Known history of recurrent miscarriage; 10)Chromosomal karyotype abnormalities in either spouse; 11)Genetic disorders that make either spouse unsuitable for childbirth as specified in the Maternal and Child Health Law;12)exposure of either spouse to teratogenic amounts of radiation, toxins, and drugs; 13)Participation in another drug or medical device clinical trial within 3 months before enrollment;14)Any medical condition/combined surgery/ medication/other clinically significant abnormal laboratory tests that, in the judgment of the investigator, may affect the outcome of the trial; 15)Known refusal or inability to comply with protocol requirements for any reason (including planned clinical visits and examinations).

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
American Fertility Association(AFS) score (mild:1-4，moderate：5-8，severe：9-12） | 3 months
  American Fertility Association(AFS) scoring performed hysteroscopically

SECONDARY OUTCOMES:
Endometrial thickness | 3 months
  Endometrial thickness measured by ultrasonography